CLINICAL TRIAL: NCT05617989
Title: Role of Non-invasive Mechanical Ventilation and Diuretics in Improving Weaning Outcome of Patients With High Lung Ultrasound Score
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mona Ammar, Assistant Professor, Ain Shams University
Other Study IDs: MD 243/2020
Record Dates: First submitted 2022-11-03; First posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Weaning Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: lung ultrasound — non-invasive ventilation and diuretic

SUMMARY:
patients who succeeded in SBT with high lung scores by ultrasound, non-invasive ventilation, and diuretic may have a role.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 21 years of age
* mechanical ventilation for more than 48 hrs
* patients successfully passed according to the traditional weaning criteria
* lung ultrasound score ≥ 17.

Exclusion Criteria:

* Significant obstructive lung diseases
* Obstructive sleep apnea
* Interstitial lung disease
* Neuromuscular disorders

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: mechanical ventilated more than 48 h with high lung score
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2021-12-04 (Actual); Study Completion 2022-04-10 (Actual)

PRIMARY OUTCOMES:
weaning failure ( number of patients) | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Medicine Ain Shams University, Cairo, Egypt